CLINICAL TRIAL: NCT06131229
Title: Emotional Education Program for the Promotion and Prevention of Mental Health in 2nd, 3rd and 4th Grade Primary School Students (ULERTUZ)
Brief Title: Two Tutorial Action Programs, Incidental and Structured, on the General Welfare of Elementary School Students.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: OIHANA SAGASTI ARRIEN (Other)
Collaborators: Universidad Nacional de Educación a Distancia (Other)
Responsible Party: Sponsor-Investigator, OIHANA SAGASTI ARRIEN, Ph.D candidate in health psychology, Oihana Sagasti
Organization: Oihana Sagasti (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: OSA-16054158C-23
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Mental Health Wellness 1
Keywords: Emotional education, tutorial action, primary school
MeSH Terms: interventions — Urination

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial of three experimental groups and three control groups is proposed, with pretest, posttest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured emotional education program (PEE) (Experimental): A tutorial action focused on a structured program of emotional education with 20 activities divided into 5 blocks with specific objectives. The program involves 34 hours of group work, one per week in the tutoring hour, throughout the 23-24 school year.
  Interventions: Behavioral: Structured emotional education program (PEE)
- Incidental tutorial action based on the school's regular curriculum (PCO) (Active Comparator): An incidental tutorial action focused on the ordinary school curriculum for the 23-24 school year.
  Interventions: Behavioral: Incidental tutorial action based on the school's regular curriculum (PCO)

INTERVENTIONS:
Behavioral: Structured emotional education program (PEE) — The principal investigator, together with the class-tutor of the experimental groups, conducts the 20 activities of which the program is composed during the hour dedicated to tutorial action. The sessions are held at Lauro School on Monday mornings in the respective classrooms, with the possibility of using the courtyard and other multipurpose rooms if the activities so require. Each session lasts one hour and is held throughout the school year 23-24.
  Arms: Structured emotional education program (PEE)
Behavioral: Incidental tutorial action based on the school's regular curriculum (PCO) — One hour tutorial action per week according to the regular school curriculum. This curriculum contemplates the incidental approach to the problems that arise in daily life and the work with the KIVA program.
  Arms: Incidental tutorial action based on the school's regular curriculum (PCO)

SUMMARY:
The aim of this paper is twofold: on the one hand, to test the effectiveness of a structured emotional education program in second, third and fourth grade primary school students and, on the other hand, to test the differential effect of such a program in relation to an incidental tutorial action focused on the ordinary school curriculum. A randomized controlled trial is proposed in Lauro Ikastola with three experimental groups (second, third and fourth of primary education) and three active control groups (one for each of the three courses) with pretest and posttest and with the duration of a school year.

DETAILED DESCRIPTION:
The implementation of emotional education in educational centers is increasingly necessary for the promotion of a complete state of physical, mental and social well-being in children throughout the entire educational stage, and especially in early stages of development.

The present work aims at a double verification. On the one hand, it is intended to test the effectiveness of a structured program of emotional education in second, third and fourth grade of primary education and, on the other hand, to test the differential effect of this program in relation to an incidental tutorial action based on the ordinary school curriculum. A randomized controlled trial is proposed in Lauro Ikastola with three experimental groups (second, third and fourth year of primary education) and three active control groups (one for each of the three courses) with pretest and posttest and with the duration of a school year.

The general objective of the proposal is the promotion of the emotional well-being of children in a particularly turbulent stage of the school cycle (2nd, 3rd and 4th grades of Primary Education) and the prevention of behavioral and/or emotional problems that may arise in later stages. The specific objectives to be achieved through the intervention in the priority population are the improvement in the following aspects: 1) Emotional intelligence; 2) Self-concept; 3) Socialization; 4) Emotional problems (depression and anxiety); 5) Behavioral problems (anger control, behavioral problems and impulsivity); and 6) Contextual problems (problems among peers). Additionally, the following two objectives are set as indirect results of the intervention in the agents involved: 5) to improve the emotional development of the parents whose children participate in the program; 6) to improve the emotional development of the tutors in charge of implementing the program.

The total sample is made up of 157 primary school students from Lauro Ikastola HLBHIP, a private school for infant, primary, secondary and high school education (municipality of Lujua, Vizcaya). From each of the three grades for which the program is intended (2nd, 3rd and 4th), two classes per grade will be selected by accessibility, which will be randomly assigned to the control group (CG) or the experimental group (GE). The emotional education program (ULERTUZ) will be applied to the experimental group and the control group will follow the academic curriculum provided by each school for each school year. The main measurement instruments will be the Adult Emotional Development Questionnaire (CDE-A), the Bar-On Emotional Intelligence Inventory EQ-I:YV, the Socialization Battery (BAS 1-2), the System for the Assessment of Children and Adolescents (SENA) and the Beck Inventory for Children and Adolescents-2 (BYI-2).

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 to 10 years.
* To be enrolled in Lauro School.
* To be in second, third or fourth grade of elementary school.

Exclusion Criteria:

* Any physical or psychological condition incompatible with the intervention

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-06-21 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Change in emotional intelligence | Baseline 1 week before treatment, Post-treatment 8 months from baseline
  Bar-On EQ-I:YV. BarOn Emotional Intelligence Inventory: youth version. Spanish version Age of application: 7 to 18 years old. The inventory is composed of 60 items to assess emotional intelligence and its different socioemotional components by means of several scales (Intrapersonal, Interpersonal, Adaptability, Stress Management and General Mood), in addition to providing an index of total Emotional Intelligence. It has two response control scales (Inconsistencies and Positive Impression), can be applied in individual or group format and lasts approximately 20-25 minutes.
Change in self-concept | Baseline 1 week before treatment, Post-treatment 8 months from baseline
  BYI-2, Beck Inventories for Children and Adolescents-2. Spanish adaptation. The Beck Child and Adolescent Inventories-2 (BYI-2) are five questionnaires published by Pearson and aimed at the assessment of depression, anxiety, anger, disruptive behavior, and self-concept in children and adolescents aged 7 to 18 years and 11 months. They are short, self-administered questionnaires that can be used separately or combined, and are simple and quick to administer. Each inventory consists of 20 statements, formulated in the first person, about thoughts, feelings or behaviors related to emotional and social disorders, to be answered with a frequency scale of four options (Never = 0; Sometimes = 1; Often = 2; Always = 3). The application time is between 5 and 10 minutes for each inventory. In the present case, we will only use the Beck Self-Concept Inventory for Children and Adolescents (BSCI-Y).

SECONDARY OUTCOMES:
Change in in emotional problems: anxiety and depression. | Baseline 1 week before treatment, Post-treatment 8 months from baseline
  SENA. Child and Adolescent Assessment System (Fernández-Pinto, I., Santamaría, P., Sánchez-Sánchez, F., Carrasco, M. A. and del Barrio, V. 2015). The purpose of the SENA is the multi-source assessment of a broad spectrum of emotional and behavioral problems (depression, anxiety, hyperactivity and impulsivity, disruptive behavior, substance use, eating behavior problems, learning problems...), contextual problems (problems with family, school and peers), as well as areas of vulnerability (emotional regulation problems, isolation, rigidity...) and psychological resources (self-esteem, social integration and competence, emotional intelligence...). The age of application is from 3 to 18 years old and has 3 different levels depending on the age of the persons assessed .
Change in behavioral problems: anger management, conduct problems and hyperactivity-impulsivity. | Baseline 1 week before treatment, Post-treatment 8 months from baseline
  SENA. Child and Adolescent Assessment System (Fernández-Pinto, I., Santamaría, P., Sánchez-Sánchez, F., Carrasco, M. A. and del Barrio, V. 2015). The purpose of the SENA is the multi-source assessment of a broad spectrum of emotional and behavioral problems (depression, anxiety, hyperactivity and impulsivity, disruptive behavior, substance use, eating behavior problems, learning problems...), contextual problems (problems with family, school and peers), as well as areas of vulnerability (emotional regulation problems, isolation, rigidity...) and psychological resources (self-esteem, social integration and competence, emotional intelligence...). The age of application is from 3 to 18 years old and has 3 different levels depending on the age of the persons assessed .
Change in contextual problems: problems with peers. | Baseline 1 week before treatment, Post-treatment 8 months from baseline
  SENA. Child and Adolescent Assessment System (Fernández-Pinto, I., Santamaría, P., Sánchez-Sánchez, F., Carrasco, M. A. and del Barrio, V. 2015). The purpose of the SENA is the multi-source assessment of a broad spectrum of emotional and behavioral problems (depression, anxiety, hyperactivity and impulsivity, disruptive behavior, substance use, eating behavior problems, learning problems...), contextual problems (problems with family, school and peers), as well as areas of vulnerability (emotional regulation problems, isolation, rigidity...) and psychological resources (self-esteem, social integration and competence, emotional intelligence...). The age of application is from 3 to 18 years old and has 3 different levels depending on the age of the persons assessed .
Change in socialization | Baseline 1 week before treatment, Post-treatment 8 months from baseline
  BAS. Socialization Battery (Silva and Martorell, 1983). Version for teachers (BAS-1) and version for parents (BAS-2). Age of application: 6 to 15 years old. These are rating scales in four facilitating dimensions of socialization (Leadership, Joviality, Social sensitivity and Respect-self-control), three disturbing ones (Aggressiveness-tertiality, Apathy-withdrawal and Anxiety-timidity) and a global scale of social adaptation or criterion-socialization. The BAS-1 (teacher compliance) has 118 items, and the BAS-2 (parent compliance) has 114 items.

CONTACTS AND LOCATIONS:
Overall Officials: OIHANA SAGASTI ARRIEN, PhDcandidate, Principal Investigator
Locations (1):
- Oihana Sagasti Arrien, Sondika, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No